CLINICAL TRIAL: NCT02794025
Title: The Effect of Esmolol on Tissue Perfusion and Clinical Prognosis of Patients With Severe Sepsis: a Prospective Cohort Study .
Brief Title: The Effect of Esmolol on Clinical Prognosis of Patients With Severe Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, the ethic committee of Fujian Provincial Hospital, Fujian Provincial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2010-001-01
Record Dates: First submitted 2016-06-04; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- esmolol group (Experimental): patients in the esmolol group received continuous infusion of esmolol via a micro-pump through a catheter placed in the superior vena cava.
  Interventions: Drug: Esmolol
- control group (Sham Comparator): Control group also received natural saline via a micro pump, in the same way the esmolol group received esmolol.
  Interventions: Drug: natural saline

INTERVENTIONS:
Drug: Esmolol — patients in the esmolol group received continuous infusion of esmolol via a micro-pump through a catheter placed in the superior vena cava. The initial dose was 0.05 mg/kg/min and was adjusted based on heart rate (HR) (target HR: 70 bpm < HR < 100 bpm within 72 hours).
  Control group also received natural saline via a micro pump, in the same way the esmolol group received esmolol.
  Other Names: β-blockers
  Arms: esmolol group
Drug: natural saline — Control group also received natural saline via a micro pump,
  Arms: control group

SUMMARY:
The purpose of this study was to investigate the effect of esmolol on hemodynamic parameters,tissue perfusion and the clinical prognosis of patients with severe sepsis

DETAILED DESCRIPTION:
enrollment:151 patients

Inclusion criteria: (1) age > 18 years; (2) severe sepsis (acute organ dysfunction secondary to infection )diagnosis according to Campaign to Save Septic Patients: 2008 Treatment Guidelines for Severe Sepsis and Septic Shock, who (3) mechanical ventilation via endotracheal intubation with a tidal volume of 6 mL/kg; and (4) satisfactory sedation and analgesic treatment, with HR > 100 bpm.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* severe sepsis (acute organ dysfunction secondary to infection )diagnosis according to Campaign to Save Septic Patients: 2008 Treatment Guidelines for Severe Sepsis and Septic Shock,
* mechanical ventilation via endotracheal intubation with a tidal volume of 6 mL/kg;
* satisfactory sedation and analgesic treatment, with HR > 100 bpm.

Exclusion Criteria:

* pre-existing cardiac dysfunction, valvular heart disease, high-degree atrioventricular block;
* acute or chronic pulmonary heart disease;
* a history of serious asthma;
* chronic renal insufficiency;
* cancer, autoimmune diseases, or contraindications for placement of deep venous catheter;
* insulin-dependent diabetes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rongguo Yu, MD, Study Director — Fujian Provincial Hospital

IPD SHARING:
Plan to Share IPD: Yes
151 patients with severe sepsis were selected and divided into the esmolol group (n = 75) or the control group (n = 76)